CLINICAL TRIAL: NCT06401499
Title: The Effect of Low Dose Pregabalin and Etoricoxib Combination on Pain in Comparison to Etoricoxib Alone in Patients Suffering From Chronic Low Back Pain
Brief Title: The Effect of Pregabalin and Etoricoxib on Pain Alone Versus in Combination
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Muhammad Ilyas (Other)
Responsible Party: Sponsor-Investigator, Muhammad Ilyas, senior lecturer, Watim Medical & Dental College
Organization: Watim Medical & Dental College (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WM&DCR/R&D(ERB)/2024/92
Record Dates: First submitted 2024-04-29; First posted 2024-05-06 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Back Pain Lower Back Chronic
MeSH Terms: interventions — Etoricoxib; Pregabalin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- etoricoxib 60mg (Experimental): tablet etoricoxib 60mg once daily for four weeks
  Interventions: Drug: etoricoxib 60mg
- pregabalin 75mg (Experimental): tablet pregabalin 75mg once daily for 4 weeks tablet etoricoxib 60mg once daily for four weeks
  Interventions: Drug: etoricoxib 60mg

INTERVENTIONS:
Drug: etoricoxib 60mg — investigator will compare effects of etoricoxib alone and in combination with pregabalin on pain relief in chronic low back pain participants
  Other Names: pregabalin 75mg

SUMMARY:
To determine the effects of pregabalin in reducing pain intensity and improving functional disability in patients with chronic low back pain of neuropathic origin when used in combination with Etoricoxib.

Hypothesis Pregabalin-etoricoxib combination is more effective than etoricoxib monotherapy in reducing pain and improving functional status in patients with chronic low back pain.

Null Hypothesis:

There is no significant difference between pregabalin-etoricoxib combination and etoricoxib monotherapy in reducing pain and improving functional status in patients with chronic low back pain.

Study Design: Comparative clinical study Setting: Watim General Hospital Duration of study: 18 months after ethical approval Sample Size: a previous study (8), was used to calculate the sample size, Using the WHO sample size calculator, a sample size of 140 patients (70 in each group) was determined with a 5% level of significance and 95% power of test.

Sampling Technique: non-probability convenience sampling. Sample selection

Inclusion criteria:

* Participants within age 20-65 years
* Both male and non-pregnant non-lactating female patients will be included in the study
* Patients experiencing CLBP symptoms from last 6 months
* No experience of previous low back surgery

Exclusion Criteria:

* Patients with the history of antidepressant, opioid, and benzodiazepine medications
* Patients with the history of CYP1A2 inhibitors usage
* Patients already taking pregabalin
* Patients with the history of suicidal ideation, severe depression, anxiety disorder psychosis, and cognitive impairment Data collection Participants will be divided into two study groups. Group A (n=70) participant will receive 60mg Etoricoxib once daily along with a placebo and Group B (n=70) participants will also receive etoricoxib 60mg once daily(15) along with a placebo for 4 weeks. At the start of week 5 the group B will start taking Pregabalin 75mg along with Etoricoxib 60mg once daily for next 4 weeks, while, group A will continue same treatment as before. At Weeks 0 and 4 and 8 of the study, participants will be evaluated. Liver enzyme levels will be measured both at the beginning and end of the trial. The pain will be measured using numeric rating scale (NRS). CLBP-related impairment will be evaluated using the self-reported 24-item Roland-Morris impairment Questionnaire (RMDQ)

DETAILED DESCRIPTION:
Introduction When back pain persists for more than three months due to a variety of non-mechanical and mechanical diseases, it is considered chronic low back pain (CLBP) Fifty percent to eighty percent of the population will have chronic low back pain (CLBP) at some time in their lives. According to a study conducted in China in 2017 "global burden of disease", CLBP affects around 4.2% of those aged 20-29, and 19.6% of people aged 30-59. The global years lived with disability for LBP were 42.5 million in 1990, and increased 52.7% to 64.9 million in 2017. In addition to being the leading cause of requesting health care services, it is also associated with substantial impairment, treatment expenditures, and sick leave. This makes it all the more important to find effective methods of treating CLBP. Treatment of CLBP remains a clinical challenge for clinicians despite the availability of several pharmacologic and non-pharmacologic techniques. The failure to address the underlying cause of the pain is a major barrier to effective treatment of CLBP. Both the nociceptive and neuropathic pain (NeP) processes may be at play in chronic low back pain, making it a disorder with a wide range of possible causes. Analysis of a US claims database found that 90% of patients with CLBP have a neuropathic component. Neuropathic pain is generally associated with more severe pain symptoms. It is the result of multiple pathways at the peripheral, spinal, and supraspinal levels that trigger pain conduction pathway changes. When compared to individuals with no neuropathic pain component, those with CLBP incur an annual treatment cost that is almost 160% greater. Therefore, it is therapeutically crucial to differentiate between the nociceptive and neuropathic processes of CLBP and to treat this illness based on its underlying mechanisms in order to improve patient outcomes and reduce disease burden.

The majority of recommendations for treating Chronic LBP are non-pharmaceutical, including multidisciplinary rehabilitation, physical therapy, acupuncture, motor control exercise, mindfulness-based stress reduction, operant therapy, low-level laser therapy, cognitive behavioral therapy, or spinal surgery. However, in cases when the patient is unresponsive , treatment is started. Etoricoxib, is a highly selective cyclooxygenase-2 (COX-2) inhibitor with anti-inflammatory, analgesic, and antipyretic properties, recommended in the relief of acute and chronic pain , Indicated for pain and inflammation in osteoarthritis, in rheumatoid arthritis, in acute gouty arthritis, in chronic low back pain. Nonsteroidal anti-inflammatory drugs and simple analgesics, only work for nociceptive pain, have poor efficacy against NeP, and have the risk of side effects with long-term use , making the treatment of CLBP even more difficult when NeP is present.

Pregabalin and gabapentin are both derived from GABA, but they have no effect on the GABAergic system. Their mechanism of action includes binding to the alpha-2/delta-1 subunit of the voltage-gated calcium channels in several areas of the central nervous system (CNS) and spinal cord, and this is sufficient to explain their analgesic, anxiolytic, and anticonvulsant pharmacological properties. Voltage-gated calcium channels are localized on presynaptic terminals, where they control neurotransmitter release. Gabapentinoids, by binding to the alpha-2/ delta-1 subunit, destabilize the macromolecular complex that keeps the calcium channel on the surface of the presynaptic terminal, promoting its internalization.

46.5 percent of Pakistanis over the age of fifty have CLBP, according to recent estimates. There was a correlation between obesity, sedentary occupations, mental health issues, inactivity, ignorance about health risks, and heavy lifting in the Pakistani population, as shown by local statistics. The incidence of this condition is greater in cities than in rural regions. In Pakistan data shows that there are studies done on other uses of pregabalin, but its role in chronic low back pain is not known to be investigated.

Rationale:

The rationale of following study is to determine the role of pregabalin in chronic low back pain in order to address neuropathic component of pain.

Data collection Participants will be divided into two study groups. Group A (n=70) participant will receive 60mg Etoricoxib once daily along with a placebo and Group B (n=70) participants will also receive etoricoxib 60mg once daily(15) along with a placebo for 4 weeks. At the start of week 5 the group B will start taking Pregabalin 75mg along with Etoricoxib 60mg once daily for next 4 weeks, while, group A will continue same treatment as before. At Weeks 0 and 4 and 8 of the study, participants will be evaluated. Liver enzyme levels will be measured both at the beginning and end of the trial. The pain will be measured using numeric rating scale (NRS). It is an 11-point scale (a lower rating suggests improvement in back pain) 0 = no pain, 1-3 = mild pain, 4- 6 = moderate pain, 7-10 = worst/severe pain. CLBP-related impairment will be evaluated using the self-reported 24-item Roland-Morris impairment Questionnaire (RMDQ), which may be scored from 0 to 24. The bigger the score, the more severe the CLBP-related disability. Patient global impression of improvement is a global index used to rate the patients' impression of their condition's response to a specific treatment. The assessment is based on the following ratings: 1 = very much better, 2 = much better, 3 = a little better, 4 = no change, 5 = a little worse, 6 = much worse, 7 = very much worse. Assessments will be performed at week 8.

Data analysis Statistical analysis was performed using SPSS for Windows version 21. Descriptive analysis will be carried out and results will be presented in frequencies alongside means and standard deviation. The data will be tested for normality using the Kolmogorov-Smirnov statistic. Independent t-tests or their non-parametric analogues (Mann-Whitney U tests) will be used to compare group means. The change in values of the variables over time will be examined using ANOVA. The confounders will be accounted for using regression models. Quantitative information will be compared using the chi-squared test (or one tailed t-test). A significance level of ≤.05 will be used.

ELIGIBILITY:
Inclusion Criteria:

* Participants within age 20-65 years
* Both male and non-pregnant non-lactating female patients will be included in the study
* Patients experiencing CLBP symptoms from last 6 months

Exclusion Criteria:

* • Patients with the history of antidepressant, opioid, and benzodiazepine medications

  * Patients with the history of CYP1A2 inhibitors usage
  * Patients already taking pregabalin
  * Patients with the history of suicidal ideation, severe depression, anxiety disorder psychosis, and cognitive impairment

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of pregabalin's effectiveness in chronic lower back will be the primary outcomes of this study | 8 weeks
  The pain will be measured using numeric rating scale (NRS). It is an 11-point scale (a lower rating suggests improvement in back pain) 0 = no pain, 1-3 = mild pain, 4- 6 = moderate pain, 7-10 = worst/severe pain. CLBP-related impairment will be evaluated using the self-reported 24-item Roland-Morris impairment Questionnaire (RMDQ), which may be scored from 0 to 24

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: atleast 3 to 6 months after study completion

REFERENCES:
- [Background] Allegri M, Montella S, Salici F, Valente A, Marchesini M, Compagnone C, Baciarello M, Manferdini ME, Fanelli G. Mechanisms of low back pain: a guide for diagnosis and therapy. F1000Res. 2016 Jun 28;5:F1000 Faculty Rev-1530. doi: 10.12688/f1000research.8105.2. eCollection 2016. PMID 27408698
- [Background] Fatoye F, Gebrye T, Odeyemi I. Real-world incidence and prevalence of low back pain using routinely collected data. Rheumatol Int. 2019 Apr;39(4):619-626. doi: 10.1007/s00296-019-04273-0. Epub 2019 Mar 8. PMID 30848349
- [Background] Wu A, March L, Zheng X, Huang J, Wang X, Zhao J, Blyth FM, Smith E, Buchbinder R, Hoy D. Global low back pain prevalence and years lived with disability from 1990 to 2017: estimates from the Global Burden of Disease Study 2017. Ann Transl Med. 2020 Mar;8(6):299. doi: 10.21037/atm.2020.02.175. PMID 32355743
- [Background] Meucci RD, Fassa AG, Faria NM. Prevalence of chronic low back pain: systematic review. Rev Saude Publica. 2015;49:1. doi: 10.1590/S0034-8910.2015049005874. Epub 2015 Oct 20. PMID 26487293
- [Background] Sakai Y, Ito K, Hida T, Ito S, Harada A. Neuropathic pain in elderly patients with chronic low back painand effects of pregabalin: a preliminary study. Asian Spine J. 2015 Apr;9(2):254-62. doi: 10.4184/asj.2015.9.2.254. Epub 2015 Apr 15. PMID 25901238
- [Background] Yeole AB, Sree Ranga Lakshmi G, Selvakumar CJ, Goni VG, Nawal CL, Valya BJ, Patel BJ, Patel RD, Pawar ED, Panigrahi R, Kumar AY, Shintre SS, Devkare PH, Dharmadhikari SK, Choudhari SY, Doshi MS, Mehta SC, Joglekar SJ. Efficacy and Safety of Pregabalin Prolonged Release-Etoricoxib Combination Compared to Etoricoxib for Chronic Low Back Pain: Phase 3, Randomized Study. Pain Ther. 2022 Dec;11(4):1451-1469. doi: 10.1007/s40122-022-00437-2. Epub 2022 Oct 12. PMID 36224489
- [Background] Caglar Okur S, Vural M, Pekin Dogan Y, Mert M, Sayiner Caglar N. The effect of pregabalin treatment on balance and gait in patients with chronic low back pain: a retrospective observational study. J Drug Assess. 2019 Feb 4;8(1):32-35. doi: 10.1080/21556660.2019.1579098. eCollection 2019. PMID 30834164
- [Background] Otto JC, Forstenpointner J, Sachau J, Hullemann P, Hukauf M, Keller T, Gierthmuhlen J, Baron R. A Novel Algorithm to Identify Predictors of Treatment Response: Tapentadol Monotherapy or Tapentadol/Pregabalin Combination Therapy in Chronic Low Back Pain? Front Neurol. 2019 Sep 13;10:979. doi: 10.3389/fneur.2019.00979. eCollection 2019. PMID 31572292
- [Background] Igarashi A, Akazawa M, Murata T, Taguchi T, Sadosky A, Ebata N, Willke R, Fujii K, Doherty J, Kobayashi M. Cost-effectiveness analysis of pregabalin for treatment of chronic low back pain in patients with accompanying lower limb pain (neuropathic component) in Japan. Clinicoecon Outcomes Res. 2015 Oct 7;7:505-20. doi: 10.2147/CEOR.S89833. eCollection 2015. PMID 26504403
- [Background] Fornasari D. Pharmacotherapy for Neuropathic Pain: A Review. Pain Ther. 2017 Dec;6(Suppl 1):25-33. doi: 10.1007/s40122-017-0091-4. Epub 2017 Nov 24. PMID 29178034
- [Background] Mathieson S, Lin CC, Underwood M, Eldabe S. Pregabalin and gabapentin for pain. BMJ. 2020 Apr 28;369:m1315. doi: 10.1136/bmj.m1315. No abstract available. PMID 32345589
- [Background] Taguchi T, Nakano S, Nozawa K. Effectiveness of Pregabalin Treatment for Neuropathic Pain in Patients with Spine Diseases: A Pooled Analysis of Two Multicenter Observational Studies in Japan. J Pain Res. 2021 Mar 16;14:757-771. doi: 10.2147/JPR.S293556. eCollection 2021. PMID 33758538
- [Background] Siddiqui AS, Javed S, Abbasi S, Baig T, Afshan G. Association Between Low Back Pain and Body Mass Index in Pakistani Population: Analysis of the Software Bank Data. Cureus. 2022 Mar 30;14(3):e23645. doi: 10.7759/cureus.23645. eCollection 2022 Mar. PMID 35510015